CLINICAL TRIAL: NCT06296706
Title: A Multicenter, Randomized, Controlled Phase III Clinical Study of Docetaxel for Injection (Albumin-bound) Versus Taxotere in Gastric Cancer
Brief Title: A Clinical Study of Docetaxel for Injection (Albumin-bound) in Patients With Gastric Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-010
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel for Injection (Albumin-bound) (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated by intravenous infusion once every 3 weeks.
  Interventions: Drug: Docetaxel for injection (Albumin-bound)
- Taxotere (Docetaxel) (Active Comparator): Taxotere will be administrated by intravenous infusion once every 3 weeks.
  Interventions: Drug: Taxotere (docetaxel)

INTERVENTIONS:
Drug: Docetaxel for injection (Albumin-bound) — Docetaxel for injection (Albumin-bound), by intravenous infusion, every 3 weeks
  Other Names: HB1801
  Arms: Docetaxel for Injection (Albumin-bound)
Drug: Taxotere (docetaxel) — Taxotere, by intravenous infusion, every 3 weeks.
  Other Names: Taxotere
  Arms: Taxotere (Docetaxel)

SUMMARY:
This trial is a multicenter, randomized, controlled phase Ш clinical study of comparison of Docetaxel for Injection (Albumin-bound) and Taxotere in locally advanced or metastatic gastric adenocarcinoma or gastroesophageal junction adenocarcinoma with previous first-line treatment failure.

DETAILED DESCRIPTION:
About 630 patients with locally advanced or metastatic gastric adenocarcinoma or gastric esophageal junction adenocarcinoma will be randomly assigned to the test group or the control group. All patients will receive Docetaxel for injection (Albumin-bound) or Taxotere for treatment until disease progression. Regular visits and imaging examinations will be conducted to compare the efficacy and safety of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-75 years (inclusive) (Whichever is on the day of signing the informed consent form).
* 2. Gastric adenocarcinoma or adenocarcinoma of gastroesophageal junction confirmed by histology or cytology.
* 3. Locally advanced or metastatic gastric adenocarcinoma or adenocarcinoma of gastroesophageal junction that has progressed after receiving first-line systematic treatment (defined as platinum/fluorouracil containing dual drug chemotherapy, with or without immunotherapy).
* 4. Evidence of disease progression on imaging during or after the last systemic treatment as confirmed by investigator.
* 5. At least one assessable lesion according to RECIST V1.1; the area should not have received previous radiotherapy, or there should be evidence of definite progress of the lesion after completion of radiotherapy.
* 6. Previous history with positive Her-2 expression requires anti-Her-2 medication; unknown Her-2 expression should define Her-2 status before enrollment.
* 7. Adequate main organ function.
* 8. Eastern Cooperative Oncology Group (ECOG) score 0-1.
* 9. Expected lifetime≥ 3 months.
* 10. Female patients of childbearing age must have a negative serum pregnancy test within 7 days prior to randomization; patients must agree to take adequate contraception from signing of ICF through 6 months after last dose, during which time women are not breastfeeding; male patients must agree to contraception and refuse sperm donation.
* 11. Fully understand this clinical trial and willing to sign a written informed consent form.

Exclusion Criteria:

* 1. Medical history of other malignant tumors or other active malignant tumors within 5 years prior to randomization (cured local tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc. can be included).
* 2. Uncontrolled serous cavity effusion requiring frequent drainage or medical intervention within 14 days before randomization (Additional intervention is required within 2 weeks after intervention, such as pleural effusion, abdominal effusion, pericardial effusion, etc., excluding exfoliative cytology testing of exudate).
* 3. Patients with central nervous system metastasis.
* 4. Patients who have used paclitaxel/docetaxel in the past (except patients with disease progression more than one year after neoadjuvant/adjuvant treatment with paclitaxel/docetaxel).
* 5. Patients whose previous medical history shows dMMR/MSI-H (deficient Mismatch Repair or High Microsatellite Instability) and who have not received immunotherapy in the past are not suitable for enrollment, and those whose dMMR/MSI status is unknown need to clarify the status before enrollment.
* 6. History of serious cardiovascular or cerebrovascular disease, including but not limited to:

  1. Serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, third degree atrioventricular block, etc;
  2. Acute coronary syndrome, congestive heart failure, stroke, or other level 3 or higher cardiovascular events occurring within 6 months before randomization;
  3. The New York Heart Association (NYHA) heart function rating of ≥ Grade Ⅱ or left ventricular ejection fraction (LVEF) of<50%;
  4. Long QTc syndrome or QTc interval>480 milliseconds, as well as the use of any known concomitant medication that can prolong the QT interval;
  5. Poor control of hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg during the screening period).
* 7. History of gastrointestinal perforation and/or fistula within 6 months before randomization.
* 8. Patients with active hepatitis B(Hepatitis B surface antigen (HBsAg) or HBcAb -positive, and in the active phase of hepatitis B (HBV-DNA ≥ 10^4 cps/mL or ≥ 2000 IU/mL)), hepatitis C(Hepatitis C antibody (Anti HCV) positive and tested positive for HCV RNA by PCR) or HIV.
* 9. Patients with severe chronic or active infections that require systemic antimicrobial, antifungal, or antiviral therapy within 14 days before randomization. Note: Patients with viral hepatitis are allowed to receive antiviral treatment.
* 10. Tuberculosis treatment history within 2 years before randomization.
* 11. Patients with gastrointestinal obstruction and active inflammatory bowel disease within 28 days before randomization.
* 12. Toxic reaction caused by any previous treatment has not recovered to level 1 or below (CTCAE5.0) (excluding anemia, alopecia, fatigue, poor appetite, or other toxicities that the investigator deems to have no safety risk to patients).
* 13. Received major organ surgery or invasive intervention treatment within 28 days before randomization. Or planned to undergo systematic or local tumor resection surgery during the study period.
* 14. Received intravenous chemotherapy or biopolymer therapy within 28 days before randomization. Or received oral chemotherapy, immunotherapy (such as interleukin, interferon, thymosin, etc.), hormone therapy, small molecule targeted therapy, or any experimental intervention within 14 days or 5 half-lives (whichever is shorter) before randomization. Received traditional Chinese medicine or traditional Chinese patent medicines with anti-tumor indications within 14 days before randomization.
* 15. Have received powerful CYP3A4 inhibitor or inducer within 14 days before randomization.
* 16. Allergic to and/or contraindication to albumin or docetaxel.
* 17. Known allergy and/or contraindication to glucocorticoids (including but not limited to active gastrointestinal ulcers, severe hypertension, severe hypokalemia, glaucoma, etc).
* 18. Patients with psychiatric neurological disorders that may affect trial adherence, or patients with a history of drug dependence/alcohol dependence.
* 19. Patients participated in another clinical study at the same time, unless it is an observational (non-intervention) clinical study or is in the follow-up period of an intervention study.
* 20. Other situations that the investigator thinks are not suitable for patients in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
OS | At the end of Cycle 1(each cycle is 21 days)
  Overall survival (OS)

SECONDARY OUTCOMES:
ORR | At the end of Cycle 1(each cycle is 21 days)
  Overall response rate (ORR)
PFS | At the end of Cycle 1(each cycle is 21 days)
  Progression-Free-Survival (PFS)
DCR | At the end of Cycle 1(each cycle is 21 days)
  Disease control rate (DCR)
DoR | At the end of Cycle 1(each cycle is 21 days)
  Duration of Response (DoR)
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | At the end of Cycle 1(each cycle is 21 days)
  The incidence and severity of adverse events (AE) and severe adverse events (SAE)
Plasma concentration of docetaxel (free and total) | At the end of Cycle 1(each cycle is 21 days)
  Plasma concentration of docetaxel (free and total)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- CSPC Zhongqi Technology(SJZ) Ltd, Shijiazhuang, Hebei, China